CLINICAL TRIAL: NCT05901506
Title: Strengthen Family Members' Understanding of Advance Care Planning With a Nurse-led, Motivational Interview Educational Intervention: A Mixed-method Feasibility Study
Brief Title: Strengthen Family Members' Understanding of Advance Care Planning With a Nurse-led, Motivational Interview
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UW 22-586
Record Dates: First submitted 2023-06-04; First posted 2023-06-13 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Family Members; Nursing Home; Older Adults
Keywords: Family Members; Advance Care Planning; Motivational Interview; Nursing Home; Older Adults
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Motivational Interview (Experimental): Participants will receive the nurse-led, motivational interview educational intervention in this group.
  Interventions: Other: a Nurse-led, Motivational Interview

INTERVENTIONS:
Other: a Nurse-led, Motivational Interview — Family member participants will receive three counselling sessions: (1) preparatory session, (2) motivation session, and (3) planning session. The preparatory session will take 10-15 minutes, and the following two sessions at weeks 2 & 3, with 30-45 min, respectively. The sessions can be delivered via face-to-face, zoom meeting, or telephones. Before each session, the nurse will first assess the family member's readiness to engage in ACP based on the State to Change algorithm. Family members who have never thought about ACP will be in the pre-contemplation state. Family members who are willing to discuss end-of-life care will be in the contemplation state. Those who are ready to talk about end-of-life planning will be in the planning state. Readiness-based ACP goals will be established, and state-matched motivational interview counseling will be customized for each participant.

SUMMARY:
The goal of this clinical trial is to strengthen the understanding of advance care planning (ACP) in family members of older adults in residential care homes with a nurse-led, motivational interview (MI) educational intervention.The main question it aims to answer is: The feasibility of the nurse-led, motivational interview educational intervention to promote family members' understanding of ACP.

Participants will receive a nurse-led, motivational interview educational intervention to see if the nurse-led, motivational interview educational intervention works in strengthening family members' knowledge on ACP and readiness for initiating conversations on ACP with their loved ones.

DETAILED DESCRIPTION:
Targeted issue: Lack of feasible method exists to empower family members of older adults in residential care homes to engage in advance care planning (ACP).

Population: Family members who are identified by a resident aged above 65 years old in residential care homes.

Intervention: A nurse-led, stage-tailored, motivational interview (MI) educational intervention.

Study aim: To evaluate the preliminary feasibility of the nurse-led, motivational interview educational intervention to promote family members' understanding of ACP.

Study method: This is a mixed-methods design, including an intervention trial and qualitative process evaluation interview. Participants will receive a nurse-led, motivational interview educational intervention and research staff will track their readiness for ACP at three-time points (before the intervention [T0], 2-week [T1], 3-week [T2] post-intervention). In addition, a post-intervention interview, regarding participants' experience of receiving the intervention, will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Identified by a resident aged above 65 years old in the residential care home as family member by the HA's definition
* Able to read and write in Chinese

Exclusion Criteria:

* Moderate to severe cognitive impairment
* Severe hearing impairment, defined as unable to participate in a telephone conversation
* Primary language other than Cantonese or Mandarin
* No access to telephone
* Cannot read or write in Chinese

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Family Members' Readiness for ACP at 2 Weeks | 2 weeks
  Family members' readiness for ACP will be measured by the researcher-developed family caregivers' ACP engagement survey (FACP-10), which consists of 10 items rated on a 5-point Likert scale. The survey assesses family caregivers' self-reported levels of ACP knowledge, readiness to discuss ACP with a loved one, self-efficacy in initiating ACP conversations with a loved one and barriers to such initiation, and emotional perceptions of and attitudes toward ACP, as well as whether having the necessary communication tools for ACP conversations. The scale scores range from 10 (the lowest) to 50 (the highest).Higher score indicates a higher readiness for ACP. Investigator developed the instrument based on the key domains reported in the Advance Care Planning Engagement Survey (ACPES) and the constructs identified in a systematic review of family caregivers' roles in ACP. The pilot data demonstrated adequate reliability of the scale in Hong Kong family caregivers.
Change from Baseline in Family Members' Readiness for ACP at 3 Weeks | 3 weeks
  Family members' readiness for ACP will be measured by the researcher-developed family caregivers' ACP engagement survey (FACP-10), which consists of 10 items rated on a 5-point Likert scale. The survey assesses family caregivers' self-reported levels of ACP knowledge, readiness to discuss ACP with a loved one, self-efficacy in initiating ACP conversations with a loved one and barriers to such initiation, and emotional perceptions of and attitudes toward ACP, as well as whether having the necessary communication tools for ACP conversations. The scale scores range from 10 (the lowest) to 50 (the highest). Higher score indicates a higher readiness for ACP. Investigator developed the instrument based on the key domains reported in the Advance Care Planning Engagement Survey (ACPES) and the constructs identified in a systematic review of family caregivers' roles in ACP. The pilot data demonstrated adequate reliability of the scale in Hong Kong family caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Chin LIN, PhD,FAAN,RN, Principal Investigator — University of Hong Kong, School of Nursing
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang T, Ho MH, Tse N, Lin CC. Motivational interviewing on engaging family members on advance care planning in residential care homes: a quasi-experimental study. BMC Nurs. 2025 Sep 26;24(1):1190. doi: 10.1186/s12912-025-03853-9. PMID 41013585